CLINICAL TRIAL: NCT05481853
Title: One Anastomosis Gastric Bypass for Severe Obesity in 6,722 Patients: Early Outcomes From the Assuta Surgery Registry
Status: Completed | Type: Observational
Sponsor: Holy Family Hospital, Nazareth, Israel (Other)
Collaborators: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Nasser Sakran, Chef Departemtn of General Surgery, Holy Family Hospital, Nazareth, Israel
Other Study IDs: 43-20-ASMC
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Morbid Obesity
Keywords: Severe obesity, Bariatric surgery, One anastomosis gastric bypass, Early postoperative complications
MeSH Terms: conditions — Obesity, Morbid; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: One Anastomosis Gastric Bypass

SUMMARY:
Background: One-anastomosis gastric bypass (OAGB) is an emerging type of bariatric metabolic surgery (BMS). Our study aimed to evaluate the short-term (≤30-day) postoperative safety of OAGB.

Methods: Electronic medical records of all OAGBs performed between January 2017 and December 2021 at a high-volume bariatric center in Israel were scanned using the MDClone software. Data regarding patients' characteristics, surgical procedure, ≤30-day postoperative complications, and their classification according to Clavien-Dindo grade were gathered. Moreover, multivariate logistic regression analysis was used to identify factors related to early postoperative complications after OAGB.

Results: A total of 6,722 patients underwent a primary (74.1%) or revisional (25.9%) OAGB procedure at our institution during the study period. Their preoperative mean age and body mass index (BMI) were 40.6±11.5 years and 41.2±4.6 kg/m2, respectively, and 75.0% were females. Respective mean operating time and length of stay were 67.3±26.6 minutes and 2.2±1.4 days. Complications occurred in 258 patients (3.8%), and include mainly bleeding (n=133, 2.0%), leaks (n=32, 0.5%), and obstruction/strictures (n=19, 0.3%). According to Clavien-Dindo classification, complication rate for grades 1-2 and grades 3a-5 were 1.6%; and 1.4%, respectively. The mortality rate was 0.03% (n=2). The rate of readmission and reoperation were 1.9% and 0.9%, respectively. Age ≥60 years, ≥3 hours of operating room time, and cholecystectomy concomitant with OAGB were independent predictors of early post-OAGB complications.

Conclusions: OAGB was found to be a safe primary and revisional BMS procedure in the ≤30-day postoperative term. The most common early complications were gastrointestinal bleeding (2.0%), leak (0.5%), and stricture (0.3%).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old, patients who received approval to undergo Bariatric and Metabolic Surgery by Assuta Medical Centers' bariatric committee, patients who have undergone primary or revisional OAGB surgery at ABCs, and patients who had complete follow-up data of 30-day post-procedure.

Exclusion Criteria: Age ≤ 18 years old

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Using the MDClone software, the electronic medical records of all patients who underwent primary or revisional OAGB at the Assuta Bariatric Centers (ABCs) between January 2017 and December 2021 were retrospectively scanned. The study was approved by the Assuta Medical Centers' ethics committee (approval number 43-20-ASMC). Informed consent was waived due to the retrospective and anonymous nature of data collected.
Sampling Method: Non-Probability Sample
Enrollment: 6722 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
≤30-day postoperative safety of OAGB based on electronic medical records of 6,722 consecutive adult patients who underwent standardized OAGB surgery at a high-volume bariatric center in Israel. | 1.1.2017 - 31/12/2021

SECONDARY OUTCOMES:
The causes and management of complications, which are potentially difficult clinical scenarios that can be faced by any bariatric surgeon. | 1.1.2017 - 31/12/2021

CONTACTS AND LOCATIONS:
Locations (1):
- Assuta Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No